CLINICAL TRIAL: NCT03885531
Title: Safety and Performance of JOURNEY™ II Cruciate Retaining (CR) Total Knee System (TKS): A Retrospective, Multicenter Study
Brief Title: Safety and Performance of JOURNEY™ II Cruciate Retaining (CR) Total Knee System (TKS)
Acronym: JIICR
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Collaborators: Nor Consult (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018.19.KNE.JIICR.RET
Record Dates: First submitted 2019-03-06; First posted 2019-03-21 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Journey II CR Total Knee System
Keywords: Journey II CR Total Knee System
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Total knee arthroplasty with Journey II CR Total Knee System — TKA with Journey II CR Total Knee System

SUMMARY:
The objective of this study is to examine the safety and performance of the Journey II CR TKS based on retrospective data.

ELIGIBILITY:
Inclusion Criteria:

* Subject received primary uni- or bilateral TKA with the Journey II CR TKS for an approved indication;
* The TKA occurred at least 12 weeks prior to enrollment

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Rheumatoid arthritis; post-traumatic arthritis, osteoarthritis or degenerative arthritis; failed osteotomies or unicompartmental replacement. This system is designed for use in patients having primary total knee replacement surgery, where the cruciate ligaments and the collateral ligaments remain intact.
Sampling Method: Non-Probability Sample
Enrollment: 586 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of adverse events reported per ISO 14155 guidelines | 7 years

SECONDARY OUTCOMES:
Length of hospital stay for primary (index) surgery | 7 years
Number of hospitalizations (admission for inpatient care) occurring after the hospitalization for the index surgery | 7 years
Length of stay of hospitalizations (admission for inpatient care) occurring after the hospitalization for the index surgery | upon occurence through 7 years of study duration
Number of rehabilitation sessions | 7 years
Duration of rehabilitation sessions in weeks | 7 years
Number and type of outpatient visits | 7 years
Number of re-operations | 7 years
Quality of Life as measured by EQ-5D-3L score | 7 years
  The EQ-5D-3L will be collected at each follow up visit. It consists of two pages - the EQ-5D descriptive system (page one) and the EQ visual analogue scale (EQ VAS) (page two). The descriptive system consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which takes one of three responses. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular dimension. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
Patient Pain Level as measured by Knee Society Score (KSS) | 7 years
  Combines an objective physician-derived component with a subjective subject-derived component. The objective section rates alignment, instability, joint motion and symptoms. Patient reported expectations and satisfaction questions evaluate pain relief, functional abilities, satisfaction and fulfillment of expectations using a subjective perspective. A functional score is derived from assessments of walking and standing, standard activities, advanced activities and discretionary activities.
Number of days before return to work | 7 years
Number of technical difficulties encountered with the device | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Navarrete, Study Chair — Smith & Nephew, Inc.
Locations (6):
- United States (6):
  - Orthopaedic Specialists of Scottsdale, Scottsdale, Arizona
  - Pikeville Medical Center, Pikeville, Kentucky
  - Reno Orthopedic Institute, Reno, Nevada
  - New York University, New York, New York
  - OrthoNeuro, New Albany, Ohio
  - Tennessee Orthopaedic Clinics, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No